CLINICAL TRIAL: NCT03913598
Title: Internet and Social Media Use in Dermatology Patients - a Survey
Brief Title: Internet and Social Media Use in Dermatology Patients
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-00009; sp19Mueller3
Record Dates: First submitted 2019-04-10; First posted 2019-04-12 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Dermatologic Diseases
Keywords: social media use; online medical services; internet use
MeSH Terms: conditions — Skin Diseases | interventions — Patient Health Questionnaire

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: patient questionnaire — self-administered patient questionnaire regarding the different aspects of internet and social media use in dermatology patients

SUMMARY:
This study is to assess Internet and social media use in dermatology patients

DETAILED DESCRIPTION:
The Internet and social media bear potential in terms of heath care consumer education, prevention of diseases and dissemination of evidence-based information. The use of the internet and social media platforms both by dermatologists and patients is rapidly evolving. In order to improve the presence and visibility of dermatology-related evidence-based informations on the Internet and in social media, the use and behavior of dermatology patients in this context is studied in more detail.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated at the Department of Dermatology of University Hospital Basel

Exclusion Criteria:

* Insufficient knowledge of German language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients treated at the Department of Dermatology of University Hospital Basel
Sampling Method: Probability Sample
Enrollment: 650 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2019-04-20 (Actual); Study Completion 2019-04-20 (Actual)

PRIMARY OUTCOMES:
Use of the Internet as a source of medical information | single time point assessment at baseline
  self-administered patient questionnaire regarding motivation to seek for medical information on the Internet
Use of Social media as a source of medical information | single time point assessment at baseline
  self-administered patient questionnaire regarding motivation to seek for medical information in Social media
Duration of Internet/ Social media use by dermatology patients | single time point assessment at baseline
  self-administered patient questionnaire covering duration of Internet/ Social media use (up to 2 hours/ day; 2 to 4 hours/day; more than 4 hours/day)
Quality assessment (by patients) of medical information provided | single time point assessment at baseline
  self-administered patient questionnaire covering quality of medical information provided on the Internet (5 point self-rating scale from very bad to very good)
Impact of internet/social media on the patient-physician relationship | single time point assessment at baseline
  self-administered patient questionnaire covering impact of internet/social media on the patient-physician relationship (self-rating scale: positive/ negative/ no impact)
Previous use of online medical services and online shopping of drugs/medications | single time point assessment at baseline
  self-administered patient questionnaire assessing previous use of online medical services and online shopping of drugs/medications (yes/ no)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Müller, Dr. med, Principal Investigator — Department of Dermatology, University Hospital Basel
Locations (1):
- Department of Dermatology, University Hospital Basel, Basel, Switzerland